CLINICAL TRIAL: NCT02499237
Title: The Effect of Zoledronic Acid Infusion in the Bone Loss Observed Following Denosumab Discontinuation in Postmenopausal Women With Low Bone Mass
Brief Title: Zoledronic Acid to Maintain Bone Mass After Denosumab Discontinuation
Acronym: AfterDmab
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: 424 General Military Hospital (Other)
Collaborators: 251 Hellenic Air Force & VA General Hospital (Other); Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Athanasios D. Anastasilakis, Consultant of Endocrinology, 424 General Military Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AfterDmab
Record Dates: First submitted 2015-07-14; First posted 2015-07-16 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Postmenopausal Osteoporosis
Keywords: osteoporosis; denosumab; zoledronic acid; bone mineral density; bone markers
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Denosumab; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Denosumab (Active Comparator): Patients with low bone mass, being treated only with denosumab in the past, who will receive another year of treatment with denosumab and subsequently discontinue treatment for one year
  Interventions: Drug: Denosumab
- Denosumab plus zoledronic acid (Experimental): Patients with low bone mass, being treated only with denosumab in the past, who will receive a single infusion of zoledronic acid and subsequently discontinue treatment for another year
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Denosumab — Treatment of low bone mass with subcutaneous injections of denosumab 60 mg every 6 months for one year
  Other Names: Prolia
  Arms: Denosumab
Drug: Zoledronic acid — Treatment of low bone mass with a single infusion of zoledronic acid 5 mg for one year
  Other Names: Aclasta
  Arms: Denosumab plus zoledronic acid

SUMMARY:
In contrast with bisphosphonates,discontinuation of denosumab results in gradual loss of bone mineral density gains. The investigators aim to evaluate whether in patients treated with denosumab, a single zoledronic acid infusion would prevent the anticipated bone loss.

DETAILED DESCRIPTION:
Discontinuation of denosumab results in a rebound rise of bone turnover markers and gradual loss of the achieved bone mineral density gains. In contrast, bisphosphonates, such as zoledronic acid, remain within the skeleton acting for several months or even years after discontinuation while maintaining bone mineral density despite the cessation of treatment. In this study, the investigators aim to evaluate changes in bone mineral density of the lumbar spine and the femoral neck, as well as in bone turnover markers one year after treatment discontinuation both in denosumab-treated women and in denosumab-treated women who switched to zoledronic acid infusion one year before treatment discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women
* osteopenic (T-score > -2.5 but < -1.0) after treatment with denosumab

Exclusion Criteria:

* secondary osteoporosis;
* diseases that could affect bone metabolism;
* medications that could affect bone metabolism;
* history of any antiosteoporotic treatment other than denosumab prior to randomization
* severe liver or kidney disease (creatinine clearance < 60ml/min/1.73m2)

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11-26 (Actual)

PRIMARY OUTCOMES:
bone mineral density of the lumbar spine | from 12 to 24 months
  differences between the 2 arms in the changes of lumbar spine bone mineral density measured by dual-energy X-ray absorptiometry

SECONDARY OUTCOMES:
bone mineral density of the femoral neck | from 12 to 24 months
  differences between the 2 arms in the changes of femoral neck bone mineral density measured by dual-energy X-ray absorptiometry
C-terminal telopeptide of type I collagen | from 12 to 15, 18, 24 months
  differences between the 2 arms in the changes of C-terminal telopeptide of type I collagen
propeptide of procollagen type I | from 12 to 15, 18, 24 months
  differences between the 2 arms in the changes of propeptide of procollagen type I
bone mineral density of the lumbar spine | from baseline to 12 months
  differences between the 2 arms in the changes of lumbar spine bone mineral density measured by dual-energy X-ray absorptiometry
bone mineral density of the femoral neck | from baseline to 12 months
  differences between the 2 arms in the changes of femoral neck bone mineral density measured by dual-energy X-ray absorptiometry

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios D Anastasilakis, PhD, Principal Investigator — 424 General Military Hospital, Thessaloniki, Greece; Polyzois Makras, PhD, Principal Investigator — 251 Airforce and VA General Hospital
Locations (2):
- Greece (2):
  - 251 Airforce & VA General Hospital, Athens
  - 424 General Military Hospital, Thessaloniki

REFERENCES:
- [Background] Miller PD, Bolognese MA, Lewiecki EM, McClung MR, Ding B, Austin M, Liu Y, San Martin J. Effect of denosumab on bone density and turnover in postmenopausal women with low bone mass after long-term continued, discontinued, and restarting of therapy: a randomized blinded phase 2 clinical trial. Bone. 2008 Aug;43(2):222-229. doi: 10.1016/j.bone.2008.04.007. Epub 2008 Apr 26. PMID 18539106
- [Background] Bone HG, Bolognese MA, Yuen CK, Kendler DL, Miller PD, Yang YC, Grazette L, San Martin J, Gallagher JC. Effects of denosumab treatment and discontinuation on bone mineral density and bone turnover markers in postmenopausal women with low bone mass. J Clin Endocrinol Metab. 2011 Apr;96(4):972-80. doi: 10.1210/jc.2010-1502. Epub 2011 Feb 2. PMID 21289258
- [Background] Black DM, Bauer DC, Schwartz AV, Cummings SR, Rosen CJ. Continuing bisphosphonate treatment for osteoporosis--for whom and for how long? N Engl J Med. 2012 May 31;366(22):2051-3. doi: 10.1056/NEJMp1202623. Epub 2012 May 9. No abstract available. PMID 22571169
- [Background] Whitaker M, Guo J, Kehoe T, Benson G. Bisphosphonates for osteoporosis--where do we go from here? N Engl J Med. 2012 May 31;366(22):2048-51. doi: 10.1056/NEJMp1202619. Epub 2012 May 9. No abstract available. PMID 22571168
- [Derived] Anastasilakis AD, Polyzos SA, Yavropoulou MP, Appelman-Dijkstra NM, Ntenti C, Mandanas S, Papatheodorou A, Makras P. Comparative Effect of Zoledronate at 6 Versus 18 Months Following Denosumab Discontinuation. Calcif Tissue Int. 2021 May;108(5):587-594. doi: 10.1007/s00223-020-00785-1. Epub 2021 Jan 2. PMID 33386953